CLINICAL TRIAL: NCT00370708
Title: Early Oral Intake Following Elective Cesarean Surgery in Iranian Women; the Economic Burdens and Patient Satisfaction
Brief Title: Early Oral Intake Following Cesarean Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1383FK
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2006-09-07 (Estimated); Status verified 2004-04

CONDITIONS: Obstetrics; Surgery
Keywords: Cesarean; Oral; Intake

INTERVENTIONS:
Procedure: Oral Intake following admittance to the postpartum ward

SUMMARY:
In this study we are trying to compare the safety and financial benefit of starting the realimentation early versus conventional oral intake following the Cesarean surgery in Iran.

DETAILED DESCRIPTION:
Cesarean delivery is announced to constitute 50% of deliveries in the Capital and 39% of all the deliveries nationwide, which is far beyond the acceptable international normal range, according to the official site of the Ministry of Health and Medical Education of the Islamic Republic of Iran [http://www.mohme.gov.ir/HNDC/Indicators/Simaye_Salamt/Simaye_Salamat.htm]. This high rate of elective cesarean deliveries might be due to several reasons which are far beyond the scope of this study. Here we tried to see whether the reduction in the time of hospitalization for these patients is safe at the expense of earlier oral realimentation and to see whether this strategy increases the patients' satisfaction or not.

ELIGIBILITY:
Inclusion Criteria:

Women who had elective cesarean deliveries under regional anesthesia

Exclusion Criteria:

1. Receiving general anesthesia, magnesium sulfate or insulin.
2. Coming across an intraoperative bowel injury.
3. Having any medical or gastrointestinal problem that prohibits early feeding

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2003-04; Study Completion 2004-02

PRIMARY OUTCOMES:
Tolerance of Oral Intake

CONTACTS AND LOCATIONS:
Overall Officials: Afsaneh Tehranian, Assist Pro, Principal Investigator — Department of Obstetrics and Gynecology, Arash Hospital, Tehran University of Medical Sciences, Tehran/Iran
Locations (1):
- Department of Obstetrics and Gynecology, Arash Hospital, Tehran, Tehran Province, Iran